CLINICAL TRIAL: NCT07231978
Title: A 2 COHORT, SINGLE DOSE, OPEN-LABEL, RANDOMIZED, PIVOTAL BIOEQUIVALENCE STUDY TO QUALIFY MANUFACTURING SITE TRANSFER FROM BARCELONETA TO ASCOLI FOR PRAZOSIN HYDROCHLORIDE CAPSULES IN HEALTHY ADULT PARTICIPANTS UNDER FASTED CONDITIONS
Brief Title: A Study to Learn How Different Forms of the Study Medicine Called Prazosin Are Taken up Into the Blood in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A0281007
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Healthy
MeSH Terms: interventions — Prazosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Participants will receive a single dose of Prazosin HCl in 4 treatments.
  Interventions: Drug: Prazosin HCl
- Cohort 2 (Experimental): Participants will receive a single dose of Prazosin HCl in 2 treatments.
  Interventions: Drug: Prazosin HCl

INTERVENTIONS:
Drug: Prazosin HCl — Administered Orally; available in capsule form
  Other Names: CP-012299

SUMMARY:
Prazosin hydrochloride (HCl) is a medicine taken by mouth that helps lower high blood pressure. It's used to treat hypertension, as well as heart failure. The purpose of this clinical trial is to prove that the prazosin HCl capsules made at the manufacturing site at Barceloneta (Puerto Rico) work the same in the body, as those made at Ascoli (Italy). This will be done by understanding how the different capsules and doses of prazosin HCL are changed and eliminated from your body after you take them. The study will also check how safe these capsules are and how well people can handle them.

This study is seeking participants ≥ 18 years old, who are healthy and have a total body weight >50 kg (110 lb). Before starting, participants will be interviewed and examined by skilled personnel to make sure they qualify. This will happen up to 28 days before the first dose of the study drug. Those who are eligible will check into the clinical research unit (CRU) the day before first dose of the study drug and stay there until 24 hours after their last dose [for approximately 9 days and 8 nights for cohort (group) 1 and 5 days and 4 nights for cohort (group) 2].

While in CRU each participant will receive by mouth either 4 capsules (cohort 1) or 2 capsules (cohort 2) of prazosin HCL at different time points. The capsules will be taken with a glass of water after overnight fasting. No food is allowed until 4 hours after taking the dose. Water is allowed freely except for 1 hour before dosing and can be consumed again 1 hour after dosing. Blood samples will be taken from participants right before they take the medicine and again after they have taken it. Electrocardiogram and blood pressure will be closely monitored.

We will compare the experiences of people receiving capsules manufactured at Barceloneta to those manufactured at Ascoli. This will help us determine if capsules from Barceloneta and Ascoli are safe and effective.

After completing all tests, participants will leave the CRU. Then, about 28 to 35 days after their final dose, they'll receive a follow-up phone call to check on their health.

The total duration of participation from the initial ("screening") visit to discharge from the CRU will be approximately 5 weeks and from the initial visit to follow up phone call will be approximately 10 weeks.

ELIGIBILITY:
Inclusion:

* Male and female participants, 18 years of age or older and who are overtly healthy as determined by medical evaluation
* Willing to comply with all study procedures
* BMI of 16-32 kg/m2; and a total body weight >50 kg (110 lb)
* Capable of giving signed informed consent

Exclusion:

* Evidence or history of clinically significant disease
* Evidence of any active suicidal ideation in the past year or suicidal behavior in the past 5 years
* Use of drugs within 14 days or 5 half-lives (whichever is longer) prior to study intervention
* Previous administration of an investigational product (drug or vaccine) within 30 days or 5 half-lives preceding the first dose of study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2026-05-04 (Estimated); Study Completion 2026-05-04 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics: Area under the plasma concentration (AUC) of prazosin | Predose, upto 5 weeks
PK: Maximum plasma concentration (Cmax) of prazosin | Predose, upto 5 weeks

SECONDARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Through study completion, approximately 10 weeks
Number of Participants With Clinical Laboratory Abnormalities | Through study completion, approximately 10 weeks
Number of participants with change from baseline in physical examinations | Through study completion, approximately 10 weeks
Number of Participants With Clinically Significant Changes From Baseline in 12-Lead Electrocardiogram (ECG) Parameters | Through study completion, approximately 10 weeks
Number of Participants With Abnormalities in Vital Signs | Through study completion, approximately 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A0281007